CLINICAL TRIAL: NCT01303835
Title: Effects of Low Dose Naltrexone on Quality of Life in High Grade Glioma Patients: A Placebo-Controlled, Double-Blind Randomized Trial
Brief Title: Low Dose Naltrexone for Glioma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Katy Peters (Other)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00027661
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-06

CONDITIONS: Malignant Glioma
Keywords: malignant glioma; glioblastoma multiforme; quality of life; naltrexone
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Experimental): Randomized patients received 4.5 mg low dose naltrexone (LDN) to be taken every night before bed.
  Interventions: Drug: LDN
- Placebo (Placebo Comparator): Randomized patients received placebo to be taken every night before bed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LDN — Randomized patients received 4.5 mg low dose naltrexone (LDN) to be taken every night before bed.
  Other Names: Low dose naltrexone; ReVia
  Arms: Naltrexone
Drug: Placebo — Randomized patients received placebo to be taken every night before bed.
  Arms: Placebo

SUMMARY:
To compare the effects of low dose naltrexone (LDN) versus placebo on quality of life in high grade glioma patients undergoing standard chemoradiation

DETAILED DESCRIPTION:
The proposed study is a placebo-controlled, randomized clinical trial. Potential participants will be identified via clinical protocol chart review of patients scheduled to attend their predetermined follow-up consultations at The Preston Robert Tisch Brain Tumor Center (PRT-BTC) at Duke University Medical Center after evaluation of treatment for newly diagnosed high grade gliomas. We will identify high grade glioma patients that will receive standard chemoradiation (radiotherapy with daily temozolomide dosed at 75 mg/m2). After obtaining written informed consent, all participants will be scheduled for baseline study assessments before starting radiotherapy. Patients will be randomized to receive either placebo or low dose naltrexone (LDN) dosed at 4.5 mg orally to be taken every evening before going to bed. Patients will be assessed at the following time points: 1. Baseline (before chemoradiation), 2. After chemoradiation (approximately 8 weeks from initial assessment), 3. Two months after standard chemoradiation (approximately 16 weeks after initial assessment), and 4. Four months after standard chemoradiation (approximately 24 weeks after initial assessment). Treatment with LDN or placebo will begin on first day of chemoradiation and will be continued for a total of 16 weeks from initial assessment. Last assessment at 24 weeks will occur 8 weeks after discontinuation of LDN or placebo. All visits will be linked to patients' clinical management visits. All testing will be performed at PRT-BTC and at Duke University Medical Center.

The following procedures will be obtained at each assessment visit:

1. Complete a six-minute walk test. The exercise test is designed to determine how far the subject can walk in six minutes. This test will take place at the PRT-BTC at Duke University Medical Center with appropriate medical supervision.
2. Blood testing that will be performed as part of each clinic visit. Approximately 10 milliliters or 2 teaspoons of blood will be drawn at each visit. This will not be additional blood work, but rather the standardized blood work that the subject will need for evaluation associated with radiation and chemotherapy treatments.

We will ask the subject to complete the following tests/questionnaires:

1. Neurocognitive testing: this testing will be performed using a computer program called CNS Vital Signs®. This program consists of verbal and visual memory tests, attention tests, reasoning tests, and speed of processing tests. The subject will use a laptop computer to complete these tests. No previous exposure to computers or computer testing is needed to complete the test.
2. Computerized Questionnaires: Four questionnaires will be presented using a computerized program. These will include Medical Outcomes Survey (MOS), Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), and Zung Self-Rating Depression Scale (ZSDS). MOS assesses general health, well-being, and quality of life. ESS asks about level of sleepiness while PSQI asks about sleep quality. Finally, ZSDS will evaluate feelings of depression and sadness.
3. Beck depression inventory (BDI): This questionnaire asks questions about the subject's levels of sadness, changes in the subject's mood, sleeping and eating patterns, the subject's level of interest in activities, thoughts and feelings the subject is having and the subject's level of concentration. This is a pen and paper questionnaire.
4. Functional Assessment of Cancer Therapy-Brain (FACT-BR) scale: This questionnaire asks questions about physical, function, emotional, and social well-being. This is a pen and paper questionnaire.
5. Functional Assessment of Cancer Therapy-Fatigue (FACIT-F) scale: This questionnaire asks questions about fatigue. This is a pen and paper questionnaire.
6. Functional Assessment of Cancer Therapy-Cognition (FACT-Cog) scale: This questionnaire asks questions about your thinking and ability to do memory, attention, and reasoning activities. This is a pen and paper questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent prior to beginning specific protocol procedures
* histologically proven high-grade glioma
* planned treatment with concurrent radiotherapy and daily oral temozolomide (with or without Avastin)
* ≥ 18 years of age
* Karnofsky performance index ≥ 70%
* must be able to ambulate unassisted for 6 minutes safely
* The Preston Robert Tisch Brain Tumor Center (PRT-BTC) neuro-oncologist's approval
* hematocrit ≥ 29%, hemoglobin ≥ 9, absolute neutrophil count (ANC) ≥ 1,500 cells/microliter, platelets ≥ 100,000 cells/microliter
* serum creatinine < 1.5 times upper limit of normal, serum glutamic oxaloacetic transaminase (SGOT) < 2.5 times upper limit of normal and bilirubin < 2.0 times upper limit of normal
* if sexually active, patients will take contraceptive measures for the duration of the treatments
* Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to administration of study drug

Exclusion Criteria:

* prior therapy with naltrexone or naloxone
* co-medication that may interfere with study results, e.g. opioids,
* known hypersensitivity to any component of naltrexone
* pregnant (positive pregnancy test) or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Peters KB, Affronti ML, Woodring S, Lipp E, Healy P, Herndon JE 2nd, Miller ES, Freeman MW, Randazzo DM, Desjardins A, Friedman HS. Effects of low-dose naltrexone on quality of life in high-grade glioma patients: a placebo-controlled, double-blind randomized trial. Support Care Cancer. 2022 Apr;30(4):3463-3471. doi: 10.1007/s00520-021-06738-0. Epub 2022 Jan 10. PMID 35001215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized to either low dose naltrexone (LDN) or placebo and were followed for 24 weeks. A patient is defined as completing the study if they completed the Quality of Life (QoL) assessments at 24 weeks.
Groups:
- Naltrexone: Randomized patients received 4.5 mg naltrexone to be taken every night before bed.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 54 | 56
Completed | 35 | 31
Not Completed | 19 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.0) | 56.7 (11.3) | 56.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Effects of Low-dose Naltrexone Versus Placebo on Change in Quality of Life (QoL) in High-grade Glioma Patients Undergoing Standard Chemoradiation From Baseline
Description: The difference in QoL scores between the 3rd QoL measurement (approximately 16 weeks from initial assessment) and the initial baseline assessment are reported. QoL instruments included are listed below. Higher scores indicate more favorable outcomes unless otherwise indicated.
  * Functional Assessment of Cancer Therapy-Brain (FACT-Br) measures general QoL reflecting symptoms associated with brain malignancies (range 0-132)
  * Functional Assessment of Chronic Illness Therapy (FACIT-F) measures level of fatigue during patients' usual daily activities (range 0-52)
  * Epworth Sleepiness Scale measures level of daytime sleepiness. Note that higher scores indicate a greater level of sleepiness (range 0-24)
  * Medical Outcomes Survey (MOS) measures QoL including physical, mental and general health via 8 domains (range 0-100 for each domain)
  * Zung Self-Rating Depression Scale quantifies the depressed status of a patient. Lower scores indicate more favorable outcome (range 20-80) A difference
Time Frame: Baseline and 16 weeks
Population: This analysis only includes those patients who completed both the initial QOL assessments and the 16 week QoL assessments, and thus number of participants may not match those reported in the participant flow module, which reports number of participants completing the trial at 24 weeks.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Low Dose Naltrexone (LDN): Randomized patients received 4.5 mg naltrexone to be taken every night before bed.
Arm/Group | Low Dose Naltrexone (LDN) | Placebo
Number analyzed (Participants) | 37 | 39
Scores on a Scale
  FACT-Brain Trial Outcome Index (TOI) | -3.73 (22.85) | -6.06 (21.72)
  FACIT-Fatigue | -4.22 (11.07) | -4.1 (13.41)
  Epworth Sleepiness Scale | 3.47 (4.37) | 0.81 (3.45)
  MOS - Physical Functioning | -5.54 (34.41) | -3.42 (29.75)
  MOS - Role Limitations due to Physical Health | 0 (51.71) | 20.39 (41.86)
  MOS - Role Limitations due to Emotional Issues | 2.69 (49.31) | 12.3 (56.11)
  MOS - Energy/Fatigue | -6.22 (29.8) | -4.61 (29.76)
  MOS - Emotional Well Being | 3.5 (21.4) | -1.89 (15.64)
  MOS - Social Functioning | 1.34 (32.38) | 7.87 (41.57)
  MOS - Pain | 10.41 (27.12) | 2.39 (24.92)
  MOS - General Health | -13.38 (17.8) | -12.11 (19.82)
  Zung Depression Scale | 0.86 (11.15) | 3.54 (8.48)

2. Secondary Outcome: Effects of Low-dose Naltrexone Versus Placebo on Change in Functional Capacity From Baseline
Description: Patients completed the 6-minute walk test (6MWT) at each QoL measurement assessment. The 6 minute walk test is a measure of functional capacity in which the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes is measured. The mean difference in distance traveled (in meters) between the 3rd QoL measurement (approximately 16 weeks from initial assessment) and the initial baseline assessment are reported. A difference greater than 0 indicates an increase in distance traveled, while a difference less than 0 indicates a decrease.
Time Frame: Baseline and 16 weeks
Population: This analysis only includes those patients who completed both the initial 6MWT assessments and the 16 week assessments, and thus number of participants may not match those reported in the participant flow module, which reports number of participants completing the trial at 24 weeks.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Low Dose Naltrexone (LDN) | Placebo
Number analyzed (Participants) | 37 | 36
Meters | 13.43 (113.7) | -6.42 (136.73)

3. Secondary Outcome: Effects of Low-dose Naltrexone Versus Placebo on Change in Neurocognitive Function From Baseline
Description: Patients completed neurocognitive testing at each QoL measurement assessment. Neurocognitive function was measured via a computerized neurocognitive test battery called CNS Vital Signs. The battery consists of 7 tests that assess verbal and visual memory, finger tapping, symbol digit coding, the Stroop Test, a test of shifting attention, and continuous performance. The battery provides scores over 9 domains with higher scores indicating better performance. Scores were normalized to a standard score mean of 100 and standard deviation of 15 using a normative sample. The mean difference in score in each domain between the 3rd QoL measurement (approximately 16 weeks from initial assessment) and the initial baseline assessment are reported. A difference greater than 0 indicates an increase in mean score, while a difference less than 0 indicates a decrease in mean score.
Time Frame: Baseline and 16 weeks
Population: This analysis only includes those patients who completed both the initial CNS Vital Signs assessments and the 16 week assessments, and thus number of participants may not match those reported in the participant flow module, which reports number of participants completing the trial at 24 weeks.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Low Dose Naltrexone (LDN) | Placebo
Number analyzed (Participants) | 21 | 25
Scores on a Scale
  Memory | -5.38 (24.03) | -0.24 (17.63)
  Processing Speed | -0.71 (24.72) | 7.32 (19.17)
  Reaction Time | -7.24 (29.61) | -8.64 (17.03)
  Verbal Memory | -0.1 (28.22) | 2 (17.29)
  Visual Memory | -8.38 (19.05) | -2.24 (19.32)
  Cognitive Flexibility | 3.62 (23.14) | 7.44 (22.12)
  Complex Attention | 7.33 (32.07) | 6.24 (18.84)
  Psychomotor Speed | -0.76 (13) | 4.72 (11.6)
  Executive Functioning | 3.9 (23.17) | 7.56 (22.87)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.4.0
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 12/54 | 17/56
Other Adverse Events (participants affected / at risk) | 51/54 | 54/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=54) | Placebo (N=56)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Edema face (General disorders) | 1 | 1
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 2 | 1
Encephalitis infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 3
Mucosal infection (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 2 | 2
White blood cell decreased (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=54) | Placebo (N=56)
Anemia (Blood and lymphatic system disorders) | 18 | 25
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Blurred vision (Eye disorders) | 2 | 5
Eye disorders - Other, specify: VISUAL FIELD CUT IN BOTH LOWER QUADRANTS (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 20 | 20
Diarrhea (Gastrointestinal disorders) | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify: CHIPPED TOOTH (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: DIVERTICULITIS (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify: DIVERTICULITIS BASELINE (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify: GI BUG (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 15 | 19
Vomiting (Gastrointestinal disorders) | 6 | 4
Chills (General disorders) | 1 | 0
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 5 | 2
Fatigue (General disorders) | 36 | 35
Fever (General disorders) | 3 | 2
Flu like symptoms (General disorders) | 1 | 0
Irritability (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Allergic reaction (Immune system disorders) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: FLU (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify: H-PYLORI (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: LLE CELLULITIS (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: LYME'S DX (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: SHINGLES (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 16 | 19
Alkaline phosphatase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 16 | 14
Blood bilirubin increased (Investigations) | 6 | 8
Creatinine increased (Investigations) | 5 | 5
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 17 | 20
Neutrophil count decreased (Investigations) | 9 | 18
Platelet count decreased (Investigations) | 29 | 31
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 5 | 2
White blood cell decreased (Investigations) | 18 | 23
Anorexia (Metabolism and nutrition disorders) | 8 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 32 | 28
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 5 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 12
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 7
Hypokalemia (Metabolism and nutrition disorders) | 15 | 10
Hyponatremia (Metabolism and nutrition disorders) | 10 | 14
Metabolism and nutrition disorders - Other, specify: PHOSPHORUS ELEVATED (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify: CRAMPS IN FEET (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: CRAMPS IN LEGS (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify: JOINT AND MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Ataxia (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 4
Dysphasia (Nervous system disorders) | 1 | 0
Edema cerebral (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 15
Hypersomnia (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 3 | 0
Nervous system disorders - Other, specify: BASELINE L HEMIPARESIS (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: DECREASED GRIP STRENGTH IN R HAND (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: GAIT DISTURBANCE (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify: L HEMIPARESIS (Nervous system disorders) | 1 | 1
Nervous system disorders - Other, specify: LE WEAKNESS (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 6 | 3
Tremor (Nervous system disorders) | 4 | 2
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 7 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 4 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Proteinuria (Renal and urinary disorders) | 3 | 5
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3
Skin and subcutaneous tissue disorders - Other, specify: DERMATITIS AT WOUND SITE (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders-MACULAR ERRYTHEMATOUS, BACK AND ABDOMEN (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No